CLINICAL TRIAL: NCT06858462
Title: Evaluation of Caries Experience Using Three Different Indices CAST, ICDAS, and WHO in a Group of Egyptian Children : a Cross-Sectional Study
Brief Title: Evaluation of Dental Caries Using Caries Assessment Spectrum and Treatment Need (CAST) Index, International Caries Detection and Assessment System (ICDAS) Index and World Health Organization (WHO) Index
Acronym: CAST/ICDAS/WHO
Status: Not yet recruiting | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Sajda Khatir Mohamed Tobai, Principal Investigator, Cairo University
Other Study IDs: Caries in three indices
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Caries Experience

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This study goals is to compare the three indices in Egyptian children aged 4 to 6 years in caries detection and time needed for the assessments which will contribute to valuable data for pediatric oral health assessments both locally and globally.

DETAILED DESCRIPTION:
This study will ensure that patients receive precise evaluations and guide early, appropriate preventive measures or treatments. Over time, this will contribute to reducing caries progression and related complications.

Also, Parents become more aware of their children's dental health status, emphasizing the importance of early detection and intervention.Furthermore , Comparing the indices will provide insights into which tool is most efficient and reliable for detecting caries in preschool children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-6 years.
* Written consent from parents or guardians for participation.
* Children who are cooperative during clinical examinations.

Exclusion Criteria:

* Children with systemic and mental diseases that might affect dental health.
* Teeth with developmental anomalies that interfere with caries assessment.
* Teeth with extensive restorations.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include children aged 4 to 6 years. They will be selected from the outpatient clinic of Pediatric Dentistry Department of the Faculty of Oral and Dental Medicine, Cairo University, according to the Eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Dental Caries Experience | Baseline ( single visit)
  The presence of dental caries will be assessed using the CAST, ICDAS, and WHO indices. The findings will provide a comparative evaluation of these indices in Egyptian children aged 4 to 6 years

SECONDARY OUTCOMES:
Time For index Application | Baseline (single visit)
  The time required to apply each caries assessment index (CAST, ICDAS, and WHO) will be measured in seconds for each child during the clinical examination

REFERENCES:
- [Background] Pauli LA, Costa VPPD, Azevedo MS, Leal SC, Goettems ML. Discriminant validity of the CAST instrument compared to the dmf index in the deciduous dentition: a cross sectional study. Braz Oral Res. 2021 Jun 16;35:e078. doi: 10.1590/1807-3107bor-2021.vol35.0078. eCollection 2021. PMID 34161415
- [Background] Attia D, ElKashlan MK, Saleh SM. Early childhood caries risk indicators among preschool children in rural Egypt: a case control study. BMC Oral Health. 2024 Jan 3;24(1):10. doi: 10.1186/s12903-023-03771-9. PMID 38172841